CLINICAL TRIAL: NCT06730399
Title: The Role of Computer-assisted Cryotherapy in the Postoperative Treatment After Total Knee Arthroplasty
Brief Title: Computer-assisted Cryotherapy After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: Cryotherapy in TKA patients
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Knee
Keywords: cryotherapy; TKA; postoperative rehabilitation; pain; recovery; opioid
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cryotherapy group: Postoperative treatment using computed-assisted-cryotherapy in the first week postoperative in addition to usual care
  Interventions: Device: Computed-assisted-cryotherapy
- Control group: Postoperative treatment according to usual care

INTERVENTIONS:
Device: Computed-assisted-cryotherapy — cryotherapy device
  Groups: Cryotherapy group

SUMMARY:
The aim of this study was to investigate whether computer-assisted cryotherapy is effective in reducing postoperative pain and analgesics consumption, next to improving functional outcome and patient satisfaction after total knee arthroplasty (TKA). The hypothesis is that computer-assisted cryotherapy has positive effects on postoperative pain after TKA.

For this purpose a single-centre non-blinded trial was designed where two groups of patients were observed, a cold (cryotherapy) C-group and a regular (control) R-group. Depended on the week they were operated patients received either usual care (R-group) or computed-assesed- cryotherapy (odd or even week; week-on/week-off principle). Patients in the C-group received next to usual postoperative care computer-assisted cryotherapy for several hours a day during the first seven postoperative days (10-12 degrees Celcius).

Primary outcome was pain, monitored with the numerical rating scale for pain. Secondary outcomes were the use of opioid escape medication, function and swelling, monitored by active range of motion, timed up and go test and circumference measurements; several patient-reported outcome measures (short term 2 and 6 weeks; and longer term 6 and 12 months postoperative); and patient satisfaction, monitored by the numerical rating scale for satisfaction.

DETAILED DESCRIPTION:
The study was conducted at the Orthopaedic Surgery Department of Martini Hospital, a teaching hospital in the Netherlands. All participants gave signed informed consent before participation. Patients with end-stage OA over the age of 18 who were scheduled for a TKA were invited to participate in this study. Exclusion criteria were rheumatoid arthritis, skin or other infections, vascular disease, other comorbidities on which cooling may have a negative effect, and strong preference for one of the treatment options. Patients were randomised into one of the two groups by a week-on/week-off principle. Patients who underwent TKA surgery in an even week received additional postoperative cryotherapy (C-group), those who had the surgery in an odd week received usual postoperative care (R-group). Surgery dates were scheduled in the usual way by the planning department of the hospital. Two weeks before surgery, patients were informed by phone as to which group they were assigned to. Both groups received the usual rapid recovery (RR) care and rehabilitation program, consisting of local infiltration analgesia during surgery, compressive bandaging for 24 h after surgery, and full weight-bearing mobilisation and active range of motion exercises starting on the day of surgery. Antibiotics were given preoperatively and postoperatively. All patients received thromboembolic prophylaxis for a period of six weeks. The Smith & Nephew (Memphis, USA) posterior stabilized (PS) GENESIS II total knee system was used for the TKA.

For the CAC in the C-group, the ZAMAR ZHC-MG665A (ZAMAR, Vrsar, Croatia) was used during hospitalisation and the smaller CAC system ZAMAR ZT Cube (ZAMAR, Vrsar, Croatia) for the home situation. The CAC system was delivered to the patient's home before the day of the surgery. Both models had a touchscreen with pre-set programs, with parameters as shown in the cooling schedule. All patients received a personal cooling brace, the ZAMAR Wrap, which transferred cold onto the skin and deep tissue around the knee. Patients in the C-group were instructed to cool the operated knee during the first seven postoperative days. The schedule they received was based on a schedule used by Thijs et al. Patients were allowed to deviate from this schedule, but were asked to document the actual cooling time and temperature in a log.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a primary TKA or UKA in the Martini Hospital.
* Age ≥ 18 years

Exclusion Criteria:

* skin (or other) infections
* rheumatoid arthritis
* vascular disease
* having a strong preference for one of the two treatment options

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all
Study Population: The study population is recruited from one large peripheral hospital in the Netherlands, the Martini Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) pain score in rest | assessed at 6 weeks postoperative
  range 0-10, where a higher score indicates more pain

SECONDARY OUTCOMES:
Numeric rating scale (NRS) pain score in rest | at baseline, daily during the first 7 days, after 2 weeks, and 6 and 12 months postoperative
  range 0-10, where a higher score indicates more pain
Numeric rating scale (NRS) pain scores while loading | at baseline, daily during the first 7 days, after 2 and 6 weeks, and 6 and 12 months postoperative
  range 0-10, where a higher score indicates more pain
Opioid use | daily during the first week after surgery
  The amount of opioid use in case of excessive pain
active Range of Motion | at baseline and at 6 weeks postoperative
  in degrees
Timed Up and Go | at baseline and at 6 weeks postoperative
  In seconds. Measure of functional mobility.
Knee circumference | at baseline and at 6 weeks postoperative
  in centimeters
Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire | preoperative and 2 and 6 weeks postoperative
  Without the sports and recreation domain. Range 0-100, where a higher score indicates less symptoms.
Work, Osteoarthritis en joint-Replacement Questionnaire (WORQ) | preoperative and 2 and 6 weeks postoperative
  Measure of work ability (functioning). Range 0-100, where a higher score indicates less functional limitations.
EuroQol 5D (EQ5D) - 5 point Likert scale | preoperative and 6 and 12 months postoperative
  Index score (0-1, closer to 1 indicates better health related quality of life); visual Analogue Scale scale about the self-perceived health status (0-100, higher indicates better self-perceived health status).
Oxford knee scores | preoperative and 6 and 12 months postoperative
  Range 0-48, where a higher score indicates less symptoms.
KOOS-PS scores (Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form) | preoperative, and 6 and 12 months postoperative
  Range 0-100, where a higher score indicates less symptoms
Numeric rating scale (NRS) satisfaction | 2 and 6 weeks postoperative, and 6 and 12 months postoperative
  patient's satisfaction with the outcome after surgery at that time point, range 0-10, where a higher score indicates more satisfaction
anchor question: patient perceived change in pain | 6 and 12 months postoperative
  the degree in which a patient experiences an improvement in pain compared to baseline (7 point Likert scale: much worse, worse, slightly worse, no change, slightly better, better, much better)
anchor question: patient perceived change in functioning | 6 and 12 months postoperative
  the degree in which a patient experiences an improvement in functioning compared to baseline (7 point Likert scale: much worse, worse, slightly worse, no change, slightly better, better, much better)
Numeric rating scal (NRS) satisfaction cryotherapy | 1 week postoperative
  Only for the patients who used the Computer-assisted-cryotherapy device: patient's satisfaction with cryotherapy. Range 0-10, where a higher score indicates more satisfaction.
Complications/Serious adverse events | from baseline until 12 months postoperative
  Keep record of the complications that occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Martini Hospital, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data will be available upon reasonable written request in conjunction with appropriate data use agreement.

REFERENCES:
- [Background] Brouwers HFG, de Vries AJ, van Zuilen M, van Kouswijk HW, Brouwer RW. The role of computer-assisted cryotherapy in the postoperative treatment after total knee arthroplasty: positive effects on pain and opioid consumption. Knee Surg Sports Traumatol Arthrosc. 2022 Aug;30(8):2698-2706. doi: 10.1007/s00167-021-06568-x. Epub 2021 Apr 26. PMID 33903923
- [Background] Thijs E, Schotanus MGM, Bemelmans YFL, Kort NP. Reduced opiate use after total knee arthroplasty using computer-assisted cryotherapy. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1204-1212. doi: 10.1007/s00167-018-4962-y. Epub 2018 May 3. PMID 29725749